CLINICAL TRIAL: NCT05760768
Title: The Effect of Individualized Exercise Guidance on Pregnancy Outcome: A Prospective Randomized Controlled Trial
Brief Title: The Effect of Individualized Exercise Guidance on Pregnancy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 018
Record Dates: First submitted 2023-02-20; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2021-11

CONDITIONS: Pregnancy Outcome; Gestational Weight Gain; Mediation; Macrosomia, Fetal
MeSH Terms: conditions — Gestational Weight Gain; Negotiating; Fetal Macrosomia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized exercise guidance group (Experimental): Participants accept individualized exercise guidance. They are also managed continuously through WeChat group chat during prenatal clinical interval.
  Interventions: Behavioral: Individualized exercise guidance
- Standard clinic prenatal care (control) group (No Intervention): Participants accept regular routine prenatal care following Chinese standard.

INTERVENTIONS:
Behavioral: Individualized exercise guidance — Participants accept individualized exercise guidance. They are also managed continuously through WeChat group chat during prenatal clinical interval.
  Arms: Individualized exercise guidance group

SUMMARY:
A single center, randomized controlled trial was conducted to investigate whether individualized exercise guidance was more effective in improving pregnancy outcomes in normal pregnant women. What's more, the trial was also conducted to find out whether there is a mediating effect between prenatal exercise and pregnancy outcomes.

DETAILED DESCRIPTION:
Fetal macrosomia refers to newborns with a birth weight more than 4000 grams, which poses varying degrees of risks to the health of both mother and infant and also affects the health outcomes of future generations. Research has found that exercise can effectively reduce the incidence of macrosomia and prevent gestational diabetes mellitus, pregnancy-induced hypertension, and excessive weight gain during pregnancy. However, every pregnant woman's individual situation and exercise habits are different, and personalized guidance based on their own circumstances is necessary during pregnancy exercise. The use of intelligent devices for supervision and management is also essential. To explore the impact of personalized exercise guidance during pregnancy on macrosomia, as well as the mediating effect of weight gain during pregnancy on exercise and macrosomia, we conducted a prospective randomized controlled clinical trial. The study included pregnant women who were over 20 years old, married, singleton, in the mid-term of pregnancy, and had no contraindications for exercise during pregnancy. They were randomly divided into an individualized exercise guidance group and standard clinic prenatal care group. Both groups received routine prenatal care and did not have any special dietary recommendations. The pregnant women in the individualized exercise guidance group received regular exercise guidance from a professional teacher and were supervised and managed through a WeChat group. The main outcome indicators were the incidence of macrosomia and the total weight gain during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* With singleton pregnancy.
* Second trimester.
* No contraindications to exercise during pregnancy.
* Be able to use smart phone for chatting, read and write basic Chinese.
* Volunteer for research.

Exclusion Criteria:

* Adverse pregnancy reaction, such as abdominal pain, vaginal bleeding and so on.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
macrosomia | From date of enrollment until the date of delivery, assessed up to 28 weeks.
  Neonatal birthweight is more than 4000 grams.
gestation weight gain（GWG） | From date of enrollment until the date of delivery, assessed up to 28 weeks.
  Weight before delivery minus weight before pregnancy.

SECONDARY OUTCOMES:
postpartum weight retention（PPWR） | From date of enrollment until the date of 42 days postpartum, assessed up to 34 weeks.
  Weight at a certain point after delivery minus weight before pregnancy.
diastasis recti abdominis（RDA） | From date of enrollment until the date of 42 days postpartum, assessed up to 34 weeks.
  The separation of the left and right rectus abdominis.

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Director — Peking union medical college hosiptal
Locations (1):
- Department of ob gyn, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang X, Wang G, Liu N, Wang Y, Zhang S, Lin H, Zhu C, Liu L, Sun Y, Ma L. Mediating effect of gestational weight gain on the preventive effect of exercise during pregnancy on macrosomia: a randomized clinical trial. BMC Pregnancy Childbirth. 2024 May 22;24(1):384. doi: 10.1186/s12884-024-06527-7. PMID 38778289